CLINICAL TRIAL: NCT04005807
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of BPN-14967 in Healthy Adult Subjects
Brief Title: Safety and Tolerability of Escalating Doses of BPN-14967 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: BPN-14967-001
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (fasted condition) (Experimental): 10 mg BPN-14967 or placebo
  Interventions: Drug: BPN-14967; Drug: Placebo
- Cohort 2 (fasted condition) (Experimental): 25 mg BPN-14967 or placebo
  Interventions: Drug: BPN-14967; Drug: Placebo
- Cohort 3 (fasted condition) (Experimental): 50 mg BPN-14967 or placebo
  Interventions: Drug: BPN-14967; Drug: Placebo
- Cohort 4 (fed condition) (Experimental): 10 mg BPN-14967 or placebo
  Interventions: Drug: BPN-14967; Drug: Placebo
- Cohort 5 (high-fat fed condition) (Experimental): 10 mg BPN-14967 or placebo
  Interventions: Drug: BPN-14967; Drug: Placebo

INTERVENTIONS:
Drug: BPN-14967 — BPN-14967 oral capsules
Drug: Placebo — Oral capsules

SUMMARY:
This is single center, randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of BPN-14967 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female (not of childbearing potential), 18 to 65 years of age, inclusive, at screening.
* The subject voluntarily consents to participate in this study and
* provides written informed consent before the start of any study-specific procedures.
* The subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for outpatient visits.
* Female subjects must be of non-childbearing potential (defined as surgically sterile [i.e., had a bilateral tubal ligation, hysterectomy, or
* bilateral oophorectomy at least 6 months before the dose of study drug] or postmenopausal for at least 1 year before study drug administration confirmed by FSH test at screening).
* Male subjects must be surgically sterile (i.e., vasectomy) for at least 3 months before screening; or agree to use a condom with spermicide when sexually active with a female partner. Male subjects must also agree to refrain from sperm donation for 90 days after study drug administration.
* The subject has a body mass index (BMI) of 18 to 30 kg/m2, inclusive, at screening and weighs 50 to 100 kg (110-220 pounds), inclusive, at screening and Check-in.
* The subject is considered to be in stable health by the investigator

Exclusion Criteria

* Any significant acute or chronic medical illness including history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease
* Any recent viral or bacterial infection.
* Participated in any clinical study in last 6 weeks.
* History of significant drug allergy
* History of significant vision, ocular or retinal disorder.
* Recent surgery, blood transfusion, drug or alcohol abuse and use of tobacco or nicotine containing products in past month.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 to the last timepoint with quantifiable concentration [AUC(0-t)] | Up to Day 8
Area under the plasma concentration versus time curve from time 0 extrapolated to infinity [AUC(0-inf)] | Up to Day 8
Maximum observed plasma concentration (Cmax) | Up to Day 8
Time to maximum observed plasma concentration (Tmax) | Up to Day 8
Terminal elimination rate constant | Up to Day 8
Terminal phase half-life (t1/2) | Up to Day 8
Apparent total body clearance (CL/F) | Up to Day 8
Apparent volume of distribution (Vz/F) | Up to Day 8
Number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs leading to discontinuation | Up to Day 10
Number of participants with Clinical Laboratory Results Abnormalities | Up to Day 10
Number of participants with Vital Sign Abnormalities | Up to Day 10
Number of participants with Physical Examination Abnormalities | Up to Day 10
Number of participants with 12-lead Electrocardiogram (ECG) Abnormalities | Up to Day 10
Number of participants with changes in visual acuity | Baseline and Day 10
Number of participants with Ocular Examination Abnormalities | Up to Day 10
Number of participants with changes in color vision | Baseline and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Petrukhin, PhD, Study Director — Professor of Ophthalmic Science, Department of Ophthalmology, Columbia University Medical Center
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
After completion of the study, data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the investigators to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority of all such issues. Data are the property of the sponsor and cannot be published without their prior authorization, but data and any publication thereof will not be unduly withheld.